CLINICAL TRIAL: NCT03440502
Title: Effect of Diabetes Mellitus on Spinal Block Criteria During Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alyaa Alaa Aldin Abd Manaf, doctor, Assiut University
Other Study IDs: Diabetes and spinal block
Record Dates: First submitted 2018-02-11; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Spinal Anaesthesia
Keywords: spinal anaesthesia; cesarean section; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group.: Parturients aged 18 or older (American Society of Anesthesiologist physical status II-III parturients ASA II-III) undergoing cesarean delivery under spinal anaesthesia, singleton pregnancy, full term, elective
  Interventions: Procedure: spinal anaesthesia
- study group: The same as control group but with DM or gestational diabetes Parturients aged 18 or older (American Society of Anesthesiologist physical status II-III parturients ASA II-III) undergoing cesarean delivery under spinal anaesthesia, singleton pregnancy, full term, elective
  Interventions: Procedure: spinal anaesthesia

INTERVENTIONS:
Procedure: spinal anaesthesia — Intrathecal block under strict aseptic conditions will be performed by median approach (L3-4 or L4-5) under sitting position by anesthesiologists . 25 Gauge sprotte spinal needles and 2-3 mLof 0.5% hyperbaric bupivacaine

SUMMARY:
The current study aimed at studying the effect of DM during pregnancy on the spinal block criteria during C.S.

The primary end point of the trial is the incidence of complete failure of spinal block.

Secondary endpoint is to determine the effect of DM on the other spinal block criteria as onset and duration of block, level of spinal block, rate of regression, hemodynamic changes, doses of inotropes and incidence of complications

DETAILED DESCRIPTION:
Regional anaesthetic techniques are now the most frequently used type of anaesthetic used for caesarean deliveries. They have a better safety profile than general anaesthesia in the pregnant woman. The choice of whether to use a spinal, epidural or combined spinal-epidural technique will depend on patient and surgical factors.

Although spinal (subarachnoid or intrathecal) anaesthesia is generally regarded as one of the most reliable types of regional block methods, the possibility of failure has long been recognized.

Most experienced practitioners would consider the incidence of failure with spinal anaesthesia to be extremely low, perhaps less than 1%. However, a figure as high as 17% has been quoted from an American teaching hospital, yet most of the failures were judged to be 'avoidable Spinal anaesthesia (SA) is a frequently used anaesthetic technique, and success rates and patient satisfaction are generally high. However, there are numerous reports of failed SA (FSA), and published failure rates in large series of SA range from 0.46% to 17%. The reasons most commonly provided to explain failure are technical problems, errors of judgement with respect to pharmacological factors, such as inadequate dose of local anaesthetic (LA), and inadequate positioning of the patient. . Proposed mechanisms for inadequate block despite correct dosing and injection technique are maldistribution , variability in the anatomy of the lumbar subarachnoid space, inadvertent subdural or epidural injection, and resistance to the effects of LA.

Successful spinal anaesthesia requires the deposition of the correct dose of the correct drug in the CSF that is in free continuity with the spinal cord and cauda equina, and that there are no barriers, either physiological, biochemical or mechanical, to prevent the normal anticipated action of the drug in the spinal cord. Gestational diabetes mellitus (GDM) refers to any degree of glucose intolerance with onset or first recognition during pregnancy. It occurs in 2-9% of all pregnancies and accounts for 90% of cases of diabetes mellitus complicating pregnancy. A1C is routinely measured approximately every 3 months in individuals with diabetes to assess the mean glucose concentration. The erythrocyte life span is ∼120 days. Thus, the 3-month interval between tests of A1C reflects the mean blood glucose over the preceding weeks to months. Hence, the rate of change of A1C in pregnancy reflects the glycemic control over the past few weeks Hoppe et al. declared diabetes mellitus (DM)as a possible cause of SA failure in a case series consisting four obstetric patients.

two possible factors may be important for quality and level of SA inpatients with DM. First is neuropathy and second is possible changes in composition of CSF such as density or volume secondary to hyperglicemia in blood and CSF .So the investigators hypothesized that DM could affect the success of SA

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for control group.

* Parturients aged 18 or older (American Society of Anesthesiologist physical status II-III parturients ASA II-III) undergoing cesarean delivery under spinal anaesthesia, singleton pregnancy, full term, elective.

Inclusion criteria for study group.

* The same as control group but with DM or gestational diabetes.

Exclusion Criteria:

* Parturients taller than 180 cm or shorter than 150 cm.
* Body mass index > 45 kg/m2.
* Known anatomical anomaly such as scolyosis or kyphosis.
* Refusal of spinal anesthesia.
* Contraindications to spinal anaesthesia (allergy to local anaesthetic or a bleeding diathesis or infection at the site of injection).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturients aged 18 or older (American Society of Anesthesiologist physical status II-III parturients ASA II-III) undergoing cesarean delivery under spinal anaesthesia, singleton pregnancy, full term, elective.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of complete failure of spinal block. | two years
  effect of DM during pregnancy on the spinal block criteria during C.S the incidence of complete failure of spinal block.

SECONDARY OUTCOMES:
determine the effect of DM on the other spinal block criteria | two years
  the other spinal block criteria as duration of block

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy JH, Islas JA, Ghia JN, Turnbull C. A retrospective study of the incidence and causes of failed spinal anesthetics in a university hospital. Anesth Analg. 1985 Jul;64(7):705-10. PMID 4014732
- [Background] Steiner LA, Hauenstein L, Ruppen W, Hampl KF, Seeberger MD. Bupivacaine concentrations in lumbar cerebrospinal fluid in patients with failed spinal anaesthesia. Br J Anaesth. 2009 Jun;102(6):839-44. doi: 10.1093/bja/aep050. Epub 2009 Mar 26. PMID 19329469
- [Background] Jovanovic L, Peterson CM. The clinical utility of glycosylated hemoglobin. Am J Med. 1981 Feb;70(2):331-8. doi: 10.1016/0002-9343(81)90770-1. PMID 6781340
- [Background] Hillier TA, Vesco KK, Pedula KL, Beil TL, Whitlock EP, Pettitt DJ. Screening for gestational diabetes mellitus: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2008 May 20;148(10):766-75. doi: 10.7326/0003-4819-148-10-200805200-00009. PMID 18490689
- [Background] Jovanovic L, Pettitt DJ. Gestational diabetes mellitus. JAMA. 2001 Nov 28;286(20):2516-8. doi: 10.1001/jama.286.20.2516. No abstract available. PMID 11722247
- See also: EFFECT OF DIABETES MELLITUS ON SPINAL ANESTHESIA FAILURE — http://www.actamedicamediterranea.com/archive/2017/medica-3/effect-of-diabetes-mellitus-on-spinal-anesthesia-failure-58f8bdc7805a9